CLINICAL TRIAL: NCT06847919
Title: Exploring the Potential Benefits of High-activity Probiotic Yogurt: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Exploring the Potential Benefits of Probiotic Yogurt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WK20250207
Record Dates: First submitted 2025-02-08; First posted 2025-02-26 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Chronic Constipation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Active Comparator): Bacterial count: ≥1000 billion CFUs per bottle Take one bottle of yogurt per day for 3 weeks
  Interventions: Dietary Supplement: Probiotic yogurt group
- Placebo group (Placebo Comparator): Product name: placebo yogurt Take one bottle of yogurt per day for 3 weeks
  Interventions: Dietary Supplement: Yogurt control group

INTERVENTIONS:
Dietary Supplement: Probiotic yogurt group — The intervention phase of this study will last 3 weeks, and each participant will make 3 visits (week 0, week 1, week 3).
  Arms: Probiotic group
Dietary Supplement: Yogurt control group — The intervention phase of this study will last 3 weeks, and each participant will make 3 visits (week 0, week 1, week 3).
  Arms: Placebo group

SUMMARY:
This study aims to evaluate the effect of a high-activity probiotic yogurt on improving symptoms of chronic constipation, observing its regulatory effects on the gut microbiota and the incidence of adverse reactions in study participants over a 21-day intervention period.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the Rome IV diagnosis criteria for chronic constipation;
2. Patients who are able to understand clinical studies and are committed to complying with study requirements and procedures;
3. Age 18-65. -

Exclusion Criteria:

1. Systemic (diabetes, autoimmune diseases, cancer), gastrointestinal or liver diseases known to be associated with alterations in the gut microbiota;
2. Patients who are pregnant or lactating;
3. have taken antimicrobials, probiotics, or drugs that inhibit stomach acid or gastrointestinal motility in the past 6 weeks;
4. Patients who changed their diet type during the study;
5. Patients who are allergic or intolerant to any component of the investigational product formulation;
6. Patients with cardiovascular, cerebrovascular, liver, kidney and hematopoietic system and other serious diseases and endocrine diseases, mental patients;
7. Stop taking the tested sample or add other drugs in the middle, unable to judge the efficacy or incomplete data;
8. short-term use of objects related to the function of the test, affecting the judgment of the result;
9. have been dieting, exercising excessively, taking weight loss medications or taking medications that may affect appetite in the past 3 months;
10. Current or past excessive use of alcohol, drugs, or supplements that may cause intestinal dysfunction or interfere with the evaluation of the efficacy of the study product -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-02-25 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Constipation symptom improvement | 3 weeks
  The Bristol Stool Form Scale (BSFS) will be used to assess improvements in constipation. The BSFS is a 9-point scale ranging from 1 to 7, where higher scores indicate softer stool consistency, approaching a liquid state. The specific scoring is as follows:
  1. Separate hard lumps, like nuts (difficult to pass)
  2. Sausage-shaped but lumpy
  3. Like a sausage but with cracks on the surface
  4. Like a sausage or snake, smooth and soft
  5. Soft blobs with clear-cut edges (passed easily)
  6. Fluffy pieces with ragged edges, a mushy stool
  7. Watery, no solid pieces, entirely liquid Scores of 4, 5, and 6 are generally considered ideal, indicating smooth bowel movements without constipation.
  Therefore, higher scores (closer to 4-6) represent improved constipation symptoms, while lower scores (1-3) indicate more severe constipation.

SECONDARY OUTCOMES:
Gut microbiota composition and diversity | 3 weeks
  Evaluating the changes in the composition and diversity of the gut microbiota before and after the intake of probiotic yogurt using high-throughput sequencing technology.
Emotional state changes | 3 weeks
  Hospital Anxiety and Depression Scale (HADS) The Hospital Anxiety and Depression Scale (HADS) will be used to quantify changes in participants' emotional state during the study period. The HADS consists of two subscales: one for anxiety (HADS-A) and one for depression (HADS-D), each containing 7 items.
  Scoring Range: Each subscale is scored from 0 to 21. Interpretation: Higher scores indicate greater levels of anxiety or depression.
Emotional state changes | 3 weeks
  Depression Anxiety Stress Scales (DASS) The Depression Anxiety Stress Scales (DASS) will be used to assess changes in participants' emotional state during the study period. The DASS includes three subscales: Depression (DASS-D), Anxiety (DASS-A), and Stress (DASS-S), each containing 14 items.
  Scoring Range: Each subscale is scored from 0 to 42. Interpretation: Higher scores indicate greater levels of depression, anxiety, or stress.
Weight management impact | 3 weeks
  Assessing the impact of probiotic yogurt intake on participants' weight management by measuring body weight.

CONTACTS AND LOCATIONS:
Locations (1):
- Suzhou Ninth People's Hospital Suzhou Ninth Hospital affiliated to Soochow University, Suzhou, Jiangsu, China